CLINICAL TRIAL: NCT03620981
Title: A Phase 2/3 Multicenter, Placebo-controlled, Randomized, Double-blind, Parallel-group Comparison Trial to Evaluate the Efficacy and Safety of Brexpiprazole (OPC-34712) in the Treatment of Patients With Agitation Associated With Dementia of the Alzheimer's Type
Brief Title: Brexpiprazole for the Treatment of Patients With Agitation Associated With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-102-00088
Record Dates: First submitted 2018-08-05; First posted 2018-08-08 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-04

CONDITIONS: Agitation Associated With Dementia of the Alzheimer's Type
MeSH Terms: interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brexpiprazole, 1mg/day (Experimental): Drug: 1mg/day Once daily for 10 weeks
  Interventions: Drug: Brexpiprazole
- Brexpiprazole, 2mg/day (Experimental): Drug: 2mg/day Once daily for 10 weeks
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): Drug: Placebo (0mg/day) Once daily for 10 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Drug: 1 tablet /day Once daily for 10 weeks
  Arms: Brexpiprazole, 1mg/day; Brexpiprazole, 2mg/day
Drug: Placebo — Placebo: 1 tablet /day Once daily for 10 weeks
  Arms: Placebo

SUMMARY:
To evaluate the superiority of brexpiprazole 1 mg or 2 mg over placebo after a 10-week treatment regimen for agitation associated with dementia of the Alzheimer's type in patients who require medication, and to investigate the safety of brexpiprazole and identify the optimum dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients who satisfy both of the following diagnostic criteria:

  1. Diagnosis of "Dementia due to Alzheimer's Disease" according to DSM-5.
  2. Diagnosis of "Probable Alzheimer's Disease" according to NINCDS-ADRDA.
* Hospitalized patients or care facility patients or care at home patients
* Patients with an MMSE score of 1 to 22
* Patients who have the agitation defined according to the "Consensus provisional definition of agitation in cognitive disorders" from the International Psychogeriatric Association (IPA)

Exclusion Criteria:

* Patients who have dementia other than dementia of the Alzheimer's type
* Patients diagnosed with delirium between 30 days before the screening examination and baseline evaluation according to DSM-5.
* Patients diagnosed with any of the following disorders according to DSM-5:

  * Schizophrenia spectrum and other psychotic disorders
  * Bipolar and related disorders
  * Major depressive disorder

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jisenkai Nanko Psychiatric Institute, Shirakawa, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

REFERENCES:
- [Derived] Nakamura Y, Adachi J, Hirota N, Iba K, Sasajima C, Shimizu K, Nakai M, Takahashi K. Brexpiprazole's impacts on patients and caregivers in agitation in Alzheimer's dementia. Alzheimers Dement. 2025 Jul;21(7):e70522. doi: 10.1002/alz.70522. PMID 40717666

RESULTS

PARTICIPANT FLOW:
Groups:
- Brexpiprazole 1 mg: Participants received a brexpiprazole 0.5 mg tablet once daily for 1 week followed by a 1 mg tablet once daily for 9 weeks.
- Brexpiprazole 2 mg: Participants received a brexpiprazole 0.5 mg tablet once daily for the first week, followed by a 1 mg tablet once daily for the second week, and then, subsequently, a 2 mg tablet once daily for the following 8 weeks.
- Placebo: Participants received placebo tablet once daily for 10 weeks.
Period: Overall Study
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
Started | 112 | 149 | 149
Completed | 83 | 102 | 116
Not Completed | 29 | 47 | 33
Not completed — Adverse Event | 14 | 38 | 25
Not completed — Lack of Efficacy | 2 | 1 | 1
Not completed — Physician Decision | 7 | 4 | 4
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Legal Representative | 2 | 1 | 1
Not completed — Withdrawal by Care Giver | 2 | 0 | 1
Not completed — Non-compliance with Study Drug | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo | Total
Number analyzed (Participants) | 112 | 149 | 149 | 410
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 4 | 15
  >=65 years | 105 | 145 | 145 | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.3 (7.4) | 80.2 (6.4) | 80.3 (6.7) | 80.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 105 | 87 | 263
  Male | 41 | 44 | 62 | 147
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 112 | 149 | 149 | 410
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 112 | 149 | 149 | 410

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cohen-Manfield Agitation Inventory(CMAI) Score at 10 Weeks After Dosing.
Description: The CMAI assessed the frequency of agitated behaviors in elderly persons, such as hitting, cursing, and restlessness. It consisted of 29 items all rated on a 1 to 7 scale with 1 being the "best" rating and 7 being the "worst" rating. The minimum possible CMAI total score was 29, and the maximum possible CMAI total score was 203. A decrease in score indicated improvement in symptoms.
Time Frame: Baseline and 10 weeks first dose, on average 10 weeks
Population: The full analysis set (FAS) comprised subjects who, after randomization, have received at least 1 dose of the IMP, and from whom CMAI total scores have been obtained at baseline and at least 1 time point after initiation of the treatment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
Number analyzed (Participants) | 108 | 148 | 147
units on a scale | -11.7 (1.20) | -15.2 (1.05) | -8.0 (1.03)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2 mg/day and placebo was performed at Week 10; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-10.0 to -4.3]
Statistical Analysis 2: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1 mg/day and placebo was performed at Week 10; Test type: Superiority; p = 0.0175, Mixed Models Analysis; LS Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-6.8 to -0.7]

2. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at 10 Weeks After Dosing.
Description: The CGI-S was used to rate the severity of agitation. Scores were: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. A decrease in score indicated improvement in symptoms.
Time Frame: Baseline and 10 weeks first dose, on average 10 weeks
Population: Efficacy sample（FAS）consisted of all participants who have received at least 1 dose of the IMP and have Baseline and at least one Post-Baseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
Number analyzed (Participants) | 108 | 148 | 147
units on a scale | -1.0 (0.1) | -1.4 (0.09) | -0.6 (0.09)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2 mg/day and placebo was performed at Week 10; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.0 to -0.5]
Statistical Analysis 2: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1 mg/day and placebo was performed at Week 10; Test type: Superiority; p = 0.0083, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to -0.1]

3. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Score at 10 Weeks After Dosing.
Description: The CGI-I Scale was clinician-rated scale which assessed the total improvement of the patient's condition compared to that at baseline. Scores range from 0 to 7: 0 = Not assessed, 1= Very much improved, 2 = Much improved, 3= Minimally improved, 4= No change, 5= Minimally worse, 6= Much worse, 7= Very much worse. Higher scores indicate worse condition.
Time Frame: Baseline and 10 weeks first dose, on average 10 weeks
Population: Efficacy sample（FAS) consisted of all participants who have received at least 1 dose of the IMP and have Baseline and at least one Post-Baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
Number analyzed (Participants) | 108 | 148 | 147
units on a scale | 3.1 (1.3) | 2.6 (1.2) | 3.5 (1.4)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2 mg/day and placebo was performed at Week 10; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel Haenszel (CMH), Last observation carried forward (LOCF); Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.2 to -0.6]
Statistical Analysis 2: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1 mg/day and placebo was performed at Week 10; Test type: Superiority; p = 0.0052, Cochran-Mantel-Haenszel; CMH, LOCF; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up for up to 35 days after the final day of IMP administration, on average 19 weeks
Description: The safety analysis comprised subjects who, after randomization, have received at least 1 dose of the IMP.
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/112 | 0/149 | 0/149
Serious Adverse Events (participants affected / at risk) | 7/112 | 9/149 | 7/149
Other Adverse Events (participants affected / at risk) | 77/112 | 113/149 | 93/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 1 mg (N=112) | Brexpiprazole 2 mg (N=149) | Placebo (N=149)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac death (General disorders) | 1 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia aspiration (Infections and infestations) | 2 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 2
Psychiatric symptom (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 1 mg (N=112) | Brexpiprazole 2 mg (N=149) | Placebo (N=149)
Constipation (Gastrointestinal disorders) | 5 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 18 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1
Gait disturbance (General disorders) | 5 | 15 | 1
Oedema peripheral (General disorders) | 2 | 2 | 3
Pyrexia (General disorders) | 9 | 11 | 8
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 3
Cellulitis (Infections and infestations) | 3 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 4 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3
Urinary tract infection (Infections and infestations) | 4 | 6 | 5
COVID-19 (Infections and infestations) | 2 | 5 | 2
Fall (Injury, poisoning and procedural complications) | 9 | 14 | 9
Contusion (Injury, poisoning and procedural complications) | 9 | 9 | 19
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 5
Skin abrasion (Injury, poisoning and procedural complications) | 4 | 8 | 9
Eye contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 6 | 0
Blood prolactin increased (Investigations) | 2 | 3 | 1
Weight decreased (Investigations) | 5 | 5 | 5
Urinary occult blood positive (Investigations) | 2 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 7 | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 3
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 9 | 16 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Akathisia (Nervous system disorders) | 0 | 1 | 3
Bradykinesia (Nervous system disorders) | 8 | 20 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 3
Dyskinesia (Nervous system disorders) | 1 | 3 | 4
Dystonia (Nervous system disorders) | 7 | 4 | 1
Extrapyramidal disorder (Nervous system disorders) | 4 | 6 | 1
Headache (Nervous system disorders) | 3 | 4 | 3
Parkinsonism (Nervous system disorders) | 5 | 5 | 0
Somnolence (Nervous system disorders) | 9 | 24 | 3
Tremor (Nervous system disorders) | 5 | 6 | 3
Parkinsonian gait (Nervous system disorders) | 2 | 3 | 0
Sedation complication (Nervous system disorders) | 3 | 11 | 2
Agitation (Psychiatric disorders) | 2 | 4 | 16
Insomnia (Psychiatric disorders) | 16 | 18 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 3 | 4
Eczema (Skin and subcutaneous tissue disorders) | 4 | 2 | 4
Erythema (Skin and subcutaneous tissue disorders) | 5 | 6 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 3
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
Skin erosion (Skin and subcutaneous tissue disorders) | 2 | 5 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 | 2 | 7
Senile xerosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03620981/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT03620981/SAP_001.pdf